CLINICAL TRIAL: NCT02422186
Title: A Randomized, Double-blind, Multicenter, Active-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Intranasal Esketamine Plus an Oral Antidepressant in Elderly Subjects With Treatment-resistant Depression
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Intranasal Esketamine Plus an Oral Antidepressant in Elderly Participants With Treatment-resistant Depression
Acronym: TRANSFORM-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107129; ESKETINTRD3005 (Other: Janssen Research & Development, LLC); 2014-004588-19 (EudraCT Number)
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Depressive Disorder, Treatment-Resistant; Esketamine; Oral Antidepressant; Elderly Participants
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine; Duloxetine Hydrochloride; Antidepressive Agents; Escitalopram; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Esketamine plus Oral Antidepressant (Experimental): Participants will self-administer esketamine intranasally twice per week for 4 weeks as a flexible dose regimen in the Double-Blind Induction Phase. All participants will start with first dose (Day 1 as 28 milligram [mg]); second dose (Day 4) is either 28 or 56 mg. All subsequent doses may be 28, 56 or 84 mg. After the first dose, all dosing decisions are determined by the investigator based on efficacy and tolerability. In addition participants will simultaneously initiate a new, open-label oral antidepressant (Duloxetine, Escitalopram, Sertraline, or Venlafaxine extended release [XR]) on Day 1 that will be continued for the duration of Double-Blind Induction Phase.
  Interventions: Drug: Esketamine; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral Antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (New Antidepressant)
- Placebo plus Oral Antidepressant (Active Comparator): Participants will self-administer matching placebo, intranasally, twice per week for 4 weeks as a flexible dose regimen in Double-Blind Induction Phase using the same titration as Esketamine. In addition participants will simultaneously initiate a new, open-label oral antidepressant (Duloxetine, Escitalopram, Sertraline, or Venlafaxine XR) on Day 1 that will be continued for the duration of Double-Blind Induction Phase.
  Interventions: Drug: Placebo; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral Antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (New Antidepressant)

INTERVENTIONS:
Drug: Esketamine — All participants will start with first dose (Day 1 as 28 milligram [mg]); second dose (Day 4) is either 28 or 56 mg. All subsequent doses may be 28, 56 or 84 mg. After the first dose, all dosing decisions are determined by the investigator based on efficacy and tolerability.
  Arms: Intranasal Esketamine plus Oral Antidepressant
Drug: Placebo — Participants will self-administer matching placebo, intranasally, twice per week for 4-weeks as a flexible dose regimen in the Double-Blind Induction Phase.
  Arms: Placebo plus Oral Antidepressant
Drug: Duloxetine (Oral Antidepressant) — Duloxetine could be selected as the oral antidepressant medication by the investigator based on review of Massachusetts General Hospital -Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and relevant prior antidepressant medication information. The minimum therapeutic dose is 60 milligram per day (mg/day).
Drug: Escitalopram (Oral Antidepressant) — Escitalopram could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Escitalopram will be given at a dose of 10 mg/day throughout the Double-Blind Induction Phase. This dose (10 mg/day) is the also the minimum therapeutic dose.
Drug: Sertraline (Oral Antidepressant) — Sertraline could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Sertraline may be titrated up to a dose of 150 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 50 mg/day.
Drug: Venlafaxine Extended Release (XR) (New Antidepressant) — Venlafaxine Extended Release could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Venlafaxine Extended Release may be titrated up to a dose of 150 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 75 mg/day.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of switching elderly participants with treatment-resistant depression (TRD) from a prior antidepressant treatment (to which they have not responded) to either intranasal esketamine plus a new oral antidepressant or switching to a new oral antidepressant plus intranasal placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind (neither the researchers nor the participants know what treatment the participant is receiving), active-controlled, multicenter study (more than 1 study site) in elderly participants with TRD to assess the efficacy, safety, and tolerability of flexible doses of intranasal esketamine plus a newly initiated oral antidepressant compared with a newly initiated oral antidepressant (active comparator) plus intranasal placebo. The study will consist of 3 phases: Screening/Prospective Observational Phase (4 to 7 weeks), Double-blind induction Phase (4 weeks), Follow up Phase (2 weeks). Participants who rollover into a long-term open-label safety study will not participate in the Follow-up Phase. At the start of the Screening/Prospective observational Phase, participant must have had documented nonresponse to at least one antidepressant treatment (based on Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire [MGH-ATRQ] criteria) in the current episode of depression, and the participant is taking a different oral antidepressant treatment on the MGH-ATRQ for at least the previous 2 weeks at or above the minimum therapeutic dose. This antidepressant treatment will be discontinued prior to the double-blind induction Phase. Participants taking benzodiazepines (at dosages equal to or less than the equivalent of 6 mg/day of lorazepam) and/or permitted non-benzodiazepine sleep medications (example, zolpidem, zaleplon) during the screening/prospective observational phase can continue these medications. All participants will start with first dose (Day 1 as 28 milligram [mg]); second dose (Day 4) is either 28 or 56 mg. All subsequent doses may be 28, 56 or 84 mg. After the first dose, all dosing decisions are determined by the investigator based on efficacy and tolerability. In addition, each participant will be assigned to receive 1 of 4 oral antidepressant medications from 2 different classes of antidepressant treatments, a Selective Serotonin Reuptake Inhibitor (SSRI) (escitalopram or sertraline) or a Serotonin and Norepinephrine Reuptake Inhibitor (SNRI) [duloxetine or venlafaxine extended release (XR)], initiated on Day 1 and continued through the double-blind induction Phase. Participants will be primarily evaluated for improvement in depressive symptoms as assessed by change in Montgomery Asberg Depression Rating Scale (MADRS) total score at Week 4. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent form (ICF), participant must be a man or woman 65 years of age or older
* At the start of the Screening/prospective observational Phase, participant must meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) [if single-episode MDD, the duration must be greater than or equal to (>=) 2 years] or recurrent MDD, without psychotic features, based upon clinical assessment and confirmed by the Mini-International Neuropsychiatric Interview (MINI)
* At the start of the Screening/Prospective observational Phase, participant must have an Inventory of Depressive Symptomatology-Clinician rated (IDS-C30) total score of greater than or equal to (>=) 31
* At the start of the Screening/Prospective observational Phase, participants must have had nonresponse (less than or equal to 25% improvement) to >=1 but less than or equal to (<=) 8 oral antidepressant treatments taken at adequate dosage and for adequate duration, as assessed using the Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and documented records by medical and pharmacy/prescription records, or a letter from the treating physician, for the current episode of depression
* Participant must be taking one of the oral antidepressant treatment with nonresponse that is documented on the MGH-ATRQ at the start of the screening/prospective observational phase
* The participant's current major depressive episode, depression symptom severity (Week 1 MADRS total score greater than or equal to 24 required) and treatment response to antidepressant treatments used in the current depressive episode (retrospectively assessed) must be confirmed for participation in a clinical study based on a Site-Independent Qualification Assessment
* Participant must be medically stable on the basis of clinical laboratory tests performed in the screening/prospective observational phase

Exclusion Criteria:

* The participant's depressive symptoms have previously demonstrated nonresponse to: Esketamine or ketamine in the current major depressive episode per clinical judgment, or all of the 4 oral antidepressant treatment options available for the double-blind induction Phase (Duloxetine, Escitalopram, Sertraline, and Venlafaxine extended release [XR]) in the current major depressive episode (based on MGH-ATRQ), or an adequate course of treatment with electroconvulsive therapy (ECT) in the current major depressive episode, defined as at least 7 treatments with unilateral ECT
* Participants who has received vagal nerve stimulation (VNS) or who has received deep brain stimulation (DBS) in the current episode of depression
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychosis, bipolar or related disorders (confirmed by the MINI), obsessive compulsive disorder (current episode only), intellectual disability ( intellectual disability [DSM-5 diagnostic codes 317, 318.0, 318.1, 318.2, 315.8, and 319]), borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* Participant has homicidal ideation/intent, per the Investigator's clinical judgment, or has suicidal ideation with some intent to act within 6 months prior to the start of the Screening/prospective observational Phase, per the Investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS) and also includes history of suicidal behavior within the past year prior to start of the screening/prospective observational phase
* Participant has a history (lifetime) of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3, 4-methylenedioxy-methamphetamine (MDMA) hallucinogen-related use disorder\
* Participant has a Mini Mental State Examination (MMSE) < 25 or <22 for those participants with less than an equivalent of high school education
* Participant has neurodegenerative disorder (eg, Alzheimer's Disease, Vascular dementia, Parkinson's disease with clinical evidence of cognitive impairment) or evidence of mild cognitive impairment (MCI)
* Participant has a history of uncontrolled hypertension; current or past history of significant pulmonary insufficiency/condition;clinically significant ECG abnormalities; current or past history of seizures; clinically significant cardiovascular disorders including cerebral and cardiac vascular disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (69):
- United States (15):
  - San Diego, California
  - New Haven, Connecticut
  - Miami, Florida
  - Marietta, Georgia
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Watertown, Massachusetts
  - New York, New York
  - Staten Island, New York
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Dallas, Texas
  - Wichita Falls, Texas
  - Charlottesville, Virginia
  - Richland, Washington
- Belgium (6):
  - Aalst
  - Bruges
  - Brussels
  - Hasselt
  - Heusden-Zolder
  - Liège
- Brazil (6):
  - Belo Horizonte
  - Fortaleza
  - Rio de Janeiro
  - Santo André
  - São José do Rio Preto
  - São Paulo
- Bulgaria (4):
  - Burgas
  - Kardzhali
  - Sofia
  - Varna
- Finland (2):
  - Helsinki
  - Kuopio
- France (9):
  - Issy-les-Moulineaux
  - La Tronche
  - Nice
  - Nîmes
  - Paris
  - Poitiers
  - Toulon
  - Toulouse
  - Tours
- Lithuania (3):
  - Kaunas
  - Šilutė
  - Vilnius
- Poland (5):
  - Bełchatów
  - Bydgoszcz
  - Gdansk
  - Torun
  - Tuszyn
- South Africa (3):
  - Cape Town
  - Garsfontein
  - Pretoria
- Spain (7):
  - Badajoz
  - Bilbao
  - Madrid
  - Ourense
  - Sant Boi de Llobregat
  - Torrevieja
  - Zamora
- Sweden (6):
  - Gothenburg
  - Halmstad
  - Lund
  - Skövde
  - Solna
  - Stockholm
- United Kingdom (3):
  - Derbyshire
  - Oxford
  - Preston

REFERENCES:
- [Derived] Doty RL, Popova V, Wylie C, Fedgchin M, Daly E, Janik A, Ochs-Ross R, Lane R, Lim P, Cooper K, Melkote R, Jamieson C, Singh J, Drevets WC. Effect of Esketamine Nasal Spray on Olfactory Function and Nasal Tolerability in Patients with Treatment-Resistant Depression: Results from Four Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Studies. CNS Drugs. 2021 Jul;35(7):781-794. doi: 10.1007/s40263-021-00826-9. Epub 2021 Jul 7. PMID 34235612
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208
- [Derived] Katz EG, Hough D, Doherty T, Lane R, Singh J, Levitan B. Benefit-Risk Assessment of Esketamine Nasal Spray vs. Placebo in Treatment-Resistant Depression. Clin Pharmacol Ther. 2021 Feb;109(2):536-546. doi: 10.1002/cpt.2024. Epub 2020 Oct 13. PMID 32860422
- See also: Randomized, Double-blind, Multicenter, Active-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Intranasal Esketamine Plus an Oral Antidepressant in Elderly Subjects with Treatment-resistant Depression — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107129&attachmentIdentifier=2db249ff-4daf-4ca5-befb-bbf9adbb3653&fileName=ESKETINTRD3005_(CR107129)_Additional_results_data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 139 participants were enrolled, out of which 138 were randomized and 1 participant was excluded due to Good Clinical Practice (GCP) non-compliance.
Groups:
- Intranasal Esketamine Plus Oral Antidepressant (AD): Participants self-administered esketamine 28 milligram (mg) or 56 mg or 84 mg intranasally twice weekly for 4 weeks (Day 1, 4, 8, 11, 15, 18, 22, 25) in DB induction phase. Also, participants initiated titration schedule for open-label oral AD with one of following: [Duloxetine (30 mg/day- Week 1, 60 mg/day- Weeks 2, 3 and 4 with MDT at 30 mg/day); Escitalopram (10 mg/day- Weeks 1-4 with MDT at 5 mg/day); Sertraline (25 mg/day- Week 1, 50 mg/day- Week 2, 100 mg/day- Week 3, 150 mg/day- Week 4 with MDT of 25 mg/Day) or Venlafaxine extended release (XR) (37.5 mg/day- Week 1, 75 mg/day- Week 2, 150 mg/day- Weeks 3, 4 with MDT of 75 mg/day)] in DB induction phase. Participants who withdrew early, before end of DB induction phase, or chose not to participate in ESKETINTRD3004 (NCT02497287) long-term safety and efficacy study, and had received at least 1 dose of intranasal esketamine 28 mg or 56 mg or 84 mg plus oral AD in DB induction phase were continued to follow-up phase for 2 weeks.
- Oral AD Plus Intranasal Placebo: Participants self-administered esketamine matched placebo intranasally twice weekly for 4 weeks (Day 1, 4, 8, 11, 15, 18, 22, 25) in double-blind (DB) induction phase. Also, participants initiated titration schedule for open-label oral antidepressant (AD) with one of the following: [Duloxetine (30 mg/day-Week 1, 60 mg/day- Weeks 2, 3 and 4 with minimum dose for tolerability (MDT) at 30 mg/day); Escitalopram (10 mg/day-Weeks 1-4 with MDT at 5 mg/day); Sertraline (25 mg/day- Week 1, 50 mg/day- Week 2, 100 mg/day- Week 3, 150 mg/day-Week 4 with MDT of 25 mg/Day) or Venlafaxine XR (37.5 mg/day- Week 1, 75 mg/day- Week 2, 150 mg/day-Weeks 3, 4 with MDT of 75 mg/day)] in DB induction phase. Participants who withdrew early, before the end of DB induction phase, or chose not to participate in ESKETINTRD3004 (NCT02497287) long-term safety and efficacy study, and had received at least 1 dose of intranasal placebo plus oral AD in DB induction phase were continued to follow-up phase for 2 weeks.
Period: Double-blind Induction Phase (4 Weeks)
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Started | 72 | 66
Full Analysis Set (FAS) | 72 | 65
Safety Analysis Set | 72 | 65
Completed | 62 | 60
Not Completed | 10 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 3 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Other | 1 | 0
Period: Follow-up Phase (2 Weeks)
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Started | 12 | 3
Completed | 8 | 3
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set was defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral antidepressant medication during the double-blind induction phase.
Groups:
- Intranasal Esketamine Plus Oral Antidepressant (AD): Participants self-administered esketamine 28 milligram (mg) or 56 mg or 84 mg intranasally twice weekly for 4 weeks (Day 1, 4, 8, 11, 15, 18, 22, 25) in DB induction phase. Also, participants initiated titration schedule for open-label oral AD with one of following: [Duloxetine (30 mg/day- Week 1, 60 mg/day- Weeks 2, 3 and 4 with MDT at 30 mg/day); Escitalopram (10 mg/day- Weeks 1-4 with MDT at 5 mg/day); Sertraline (25 mg/day- Week 1, 50 mg/day- Week 2, 100 mg/day- Week 3, 150 mg/day- Week 4 with MDT of 25 mg/Day) or Venlafaxine extended release (XR) (37.5 mg/day- Week 1, 75 mg/day- Week 2, 150 mg/day- Weeks 3, 4 with MDT of 75 mg/day)] in DB induction phase. Participants who withdrew early, before end of DB induction phase, or chose not to participate in ESKETINTRD3004 (NCT02497287) long-term safety and efficacy study, and had received at least 1 dose of intranasal esketamine 28 mg or 56 mg or 84 mg+ oral AD in DB induction phase were continued to follow-up phase for 2 weeks.
- Oral AD Plus Intranasal Placebo: Participants self-administered esketamine matched placebo intranasally twice weekly for 4 weeks (Day 1, 4, 8, 11, 15, 18, 22, 25) in double-blind (DB) induction phase. Also, participants initiated titration schedule for open-label oral antidepressant (AD) with one of the following: [Duloxetine (30 mg/day- Week 1, 60 mg/day- Weeks 2, 3 and 4 with minimum dose for tolerability (MDT) at 30 mg/day); Escitalopram (10 mg/day- Weeks 1-4 with MDT at 5 mg/day); Sertraline (25 mg/day- Week 1, 50 mg/day- Week 2, 100 mg/day- Week 3, 150 mg/day- Week 4 with MDT of 25 mg/Day) or Venlafaxine XR (37.5 mg/day- Week 1, 75 mg/day- Week 2, 150 mg/day- Weeks 3, 4 with MDT of 75 mg/day)] in DB induction phase. Participants who withdrew early, before the end of DB induction phase, or chose not to participate in ESKETINTRD3004 (NCT02497287) long-term safety and efficacy study, and had received at least 1 dose of intranasal placebo+ oral AD in DB induction phase were continued to follow-up phase for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo | Total
Number analyzed (Participants) | 72 | 65 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 72 | 65 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (4.79) | 69.4 (4.15) | 70 (4.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 40 | 85
  Male | 27 | 25 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 59 | 59 | 118
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 66 | 64 | 130
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 2 | 4 | 6
  Brazil | 1 | 0 | 1
  Bulgaria | 3 | 0 | 3
  Finland | 1 | 1 | 2
  France | 4 | 3 | 7
  Italy | 6 | 3 | 9
  Lithuania | 2 | 0 | 2
  Poland | 4 | 3 | 7
  South Africa | 2 | 5 | 7
  Spain | 4 | 4 | 8
  Sweden | 8 | 6 | 14
  United Kingdom | 1 | 0 | 1
  United States | 34 | 36 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])- Mixed-Effects Model Using Repeated Measures (MMRM) Analysis
Description: The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items (to evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel [interest level], pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score range of 0-60. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline up to Endpoint (Double-blind Induction Phase[Day 28])
Population: The full analysis set (FAS) was defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral antidepressant medication during the double-blind induction phase. Here, N (Overall number of participants analyzed) signifies number of participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 63 | 60
Units on a scale | -10.0 (12.74) | -6.3 (8.86)
Statistical Analysis 1: Comparison: Intranasal Esketamine Plus Oral Antidepressant (AD) vs Oral AD Plus Intranasal Placebo; Test type: Superiority; p = 0.059, Mixed Model for Repeated Measures; Difference of Least Square (LS) Means = -3.6, 95% CI 2-sided [-7.20 to 0.07]

2. Primary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score to Endpoint (Double-blind Induction Phase [Day 28])- Analysis of Covariance (ANCOVA) Analysis
Description: The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items (to evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel [interest level], pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score range of 0-60. Higher scores represent a more severe condition. Negative change in score indicates improvement. Missing data was imputed using Last Observation Carried Forward (LOCF) method and last post baseline observation during the double-blind induction phase was carried forward as the "End Point" for that phase.
Time Frame: Baseline and Endpoint (Double-blind Induction Phase [Day 28])
Population: The full analysis set was defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral antidepressant medication during the double-blind induction phase. Here, N (Overall number of participants analyzed) signifies number of participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 71 | 64
Units on a scale | -9.3 (12.28) | -5.6 (9.11)
Statistical Analysis 1: Comparison: Intranasal Esketamine Plus Oral Antidepressant (AD) vs Oral AD Plus Intranasal Placebo; Test type: Other; p = 0.052, ANCOVA; Least Square (LS) Mean Difference = -3.6, 95% CI 2-sided [-7.16 to -0.03]

3. Secondary Outcome: Percentage of Participants Who Achieved >=50% Reduction From Baseline in MADRS Total Score at Endpoint (Double-blind Induction Phase [Day 28]) (LOCF Data)
Description: Percentage of participants with greater than or equal to (>=50) percent (%) reduction from baseline are reported. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. Missing data was imputed using LOCF method and last post baseline observation during the double-blind induction phase was carried forward as the "End Point" for that phase.
Time Frame: At Endpoint-Double-blind Induction Phase [Day 28]
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 71 | 64
Percentage of Participants | 23.9 | 12.5

4. Secondary Outcome: Percentage of Participants in Remission (MADRS<=12) at Endpoint (Double-blind Induction Phase [Day 28]) (LOCF Data)
Description: Remission was defined as participants who had a MADRS total score of less than or equal to (=<) 12. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. Missing data was imputed using LOCF method and last post baseline observation during the double-blind induction phase was carried forward as the "End Point" for that phase.
Time Frame: At Endpoint-Double-blind Induction Phase [Day 28]
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 71 | 64
Percentage of Participants | 15.5 | 6.3

5. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score to Endpoint (Double-blind Induction Phase [Day 28])- ANCOVA Analysis on Ranks
Description: CGI-S provides an overall clinician-determined summary measure of the severity of the participants illness including participants history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participants ability to function. The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. Missing data was imputed using LOCF method and last post baseline observation during the double-blind induction phase was carried forward as the "End Point" for that phase.
Time Frame: Baseline and Endpoint (Double-blind Induction Phase [Day 28])
Population: as for outcome 2
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 71 | 65
Units on a scale | -1.0 [-4 to 1] | 0.0 [-4 to 3]

6. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) to Endpoint (Double-blind Induction Phase [Day 28]): Health Status Index
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a health status index (HSI). HSI ranges from -0.148 (health state value equal to dead) and 0.949 (full health), is anchored at 0 (dead) and 1 (full health).
Time Frame: Baseline and Endpoint (Double-blind Induction Phase [Day 28])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 70 | 64
Units on a scale | 0.081 (0.2624) | 0.026 (0.2235)

7. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) to Endpoint (Double-blind Induction Phase [Day 28]): EQ-VAS
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. The EQ VAS self-rating records the respondent's own assessment of his or her overall health status at the time of completion, on a scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Time Frame: Baseline and Endpoint (Double-blind Induction Phase [Day 28])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 70 | 64
Units on a scale | 6.2 (22.78) | 4.4 (20.60)

8. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) to Endpoint (Double-blind Induction Phase [Day 28]): Sum Score
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ VAS). EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a Health Status Index (HSI). HSI ranges from -0.148 (health state value equal to dead) and 0.949 (full health). EQ VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: Baseline and Endpoint (Double-blind Induction Phase [Day 28])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine Plus Oral Antidepressant (AD) | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 70 | 64
Units on a scale | -6.6 (20.53) | -1.6 (16.21)

ADVERSE EVENTS:
Time Frame: Up to 13 weeks
Description: The population analyzed included safety analysis set- all randomized participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant medication during the double-blind induction phase and follow-up analysis set- all participants who entered the follow-up phase.
Groups:
- DB Phase: Intranasal Esketamine + Oral AD (4 Weeks): Participants self-administered esketamine 28 milligram (mg) or 56 mg or 84 mg intranasally twice weekly for 4 weeks (Day 1, 4, 8, 11, 15, 18, 22, 25) in DB induction phase. Also, participants initiated titration schedule for open-label oral AD with one of following: [Duloxetine (30 mg/day- Week 1, 60 mg/day- Weeks 2, 3 and 4 with MDT at 30 mg/day); Escitalopram (10 mg/day- Weeks 1-4 with MDT at 5 mg/day); Sertraline (25 mg/day- Week 1, 50 mg/day- Week 2, 100 mg/day- Week 3, 150 mg/day- Week 4 with MDT of 25 mg/Day) or Venlafaxine extended release (XR) (37.5 mg/day- Week 1, 75 mg/day- Week 2, 150 mg/day- Weeks 3, 4 with MDT of 75 mg/day)] in DB induction phase.
- DB Phase: Oral AD + Intranasal Placebo (4 Weeks): Participants self-administered esketamine matched placebo intranasally twice weekly for 4 weeks (Day 1, 4, 8, 11, 15, 18, 22, 25) in double-blind (DB) induction phase. Also, participants initiated titration schedule for open-label oral antidepressant (AD) with one of the following: [Duloxetine (30 mg/day- Week 1, 60 mg/day- Weeks 2, 3 and 4 with minimum dose for tolerability (MDT) at 30 mg/day); Escitalopram (10 mg/day- Weeks 1-4 with MDT at 5 mg/day); Sertraline (25 mg/day- Week 1, 50 mg/day- Week 2, 100 mg/day- Week 3, 150 mg/day- Week 4 with MDT of 25 mg/Day) or Venlafaxine XR (37.5 mg/day- Week 1, 75 mg/day- Week 2, 150 mg/day- Weeks 3, 4 with MDT of 75 mg/day)] in DB induction phase.
- Follow-up Phase: Intranasal Esketamine + Oral AD (2 Weeks): Participants who withdrew early, before end of DB induction phase, or chose not to participate in ESKETINTRD3004 (NCT02497287) long-term safety and efficacy study, and had received at least 1 dose of intranasal esketamine 28 mg or 56 mg or 84 mg+ oral AD in DB induction phase were continued to follow-up phase for 2 weeks.
- Follow-up Phase: Oral AD + Intranasal Placebo (2 Weeks): Participants who withdrew early, before the end of DB induction phase, or chose not to participate in ESKETINTRD3004 (NCT02497287) long-term safety and efficacy study, and had received at least 1 dose of intranasal placebo+ oral AD in DB induction phase were continued to follow-up phase for 2 weeks.
Arm/Group | DB Phase: Intranasal Esketamine + Oral AD (4 Weeks) | DB Phase: Oral AD + Intranasal Placebo (4 Weeks) | Follow-up Phase: Intranasal Esketamine + Oral AD (2 Weeks) | Follow-up Phase: Oral AD + Intranasal Placebo (2 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/65 | 0/12 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/72 | 2/65 | 0/12 | 0/3
Other Adverse Events (participants affected / at risk) | 44/72 | 22/65 | 1/12 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase: Intranasal Esketamine + Oral AD (4 Weeks) (N=72) | DB Phase: Oral AD + Intranasal Placebo (4 Weeks) (N=65) | Follow-up Phase: Intranasal Esketamine + Oral AD (2 Weeks) (N=12) | Follow-up Phase: Oral AD + Intranasal Placebo (2 Weeks) (N=3)
Gait Disturbance (General disorders) | 0 | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Feeling of Despair (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase: Intranasal Esketamine + Oral AD (4 Weeks) (N=72) | DB Phase: Oral AD + Intranasal Placebo (4 Weeks) (N=65) | Follow-up Phase: Intranasal Esketamine + Oral AD (2 Weeks) (N=12) | Follow-up Phase: Oral AD + Intranasal Placebo (2 Weeks) (N=3)
Vertigo (Ear and labyrinth disorders) | 8 | 2 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 0 | 1
Fatigue (General disorders) | 9 | 5 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 6 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 9 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 15 | 4 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 3 | 0 | 0
Headache (Nervous system disorders) | 9 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 4 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 5 | 0 | 0
Dissociation (Psychiatric disorders) | 9 | 1 | 0 | 0
Dysphoria (Psychiatric disorders) | 4 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will be withheld such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT02422186/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT02422186/SAP_001.pdf